CLINICAL TRIAL: NCT06224985
Title: Computational Anatomy in Surgery for Childhood Tumours and Malformations
Acronym: IMAG2
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMAG 2
Record Dates: First submitted 2024-01-03; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Malformation; Tumor; Paediatric Surgery; 3D Imaging
MeSH Terms: conditions — Congenital Abnormalities; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Malformation
- Tumors
- Controls

SUMMARY:
This study is part of the launch of a multidisciplinary project called IMAG2, for image-guided minimally invasive surgery. It involves collaboration between the radiology and surgery teams at Necker Hospital and the Image Processing and Interpretation (TII) team at the LTCI at Télécom ParisTech.

To make a decision, surgeons need access to a 3D model reflecting the anatomy of the specific patient and its pathological variations. Patient-specific 3D reconstruction provides a significant improvement, leading to a precise assessment of the malformation or tumour and its relationship with surrounding organs, nerves and vessels. It allows the surgeon to simulate a pre-operative procedure, which is a definite advantage in terms of safe, effective and curative surgery, particularly in oncology. MRI has been chosen as the basic imaging technique because of its non-irradiating nature and the current lack of 3D MRI reconstruction technology.

The study aims to provide an aid to diagnosis and surgical planning by developing dedicated methods and algorithms for segmenting not only the tumour but also the main anatomical components surrounding the tumour from 3D MRI imaging data. The imaging will be performed on a 3 Tesla MRI. The data will be that required for diagnosis and surgical planning, acquired on a routine clinical basis with an expected benefit for patients.

ELIGIBILITY:
To be included, patients must meet the following criteria:

* Patient aged between 5 months and 17 years
* Patient with a confirmed diagnosis of :

  * Abdomino-pelvic tumour
  * Pelvic malformation
* Patient whose parents or legal guardians have read, accepted and signed the study consent form
* Patients whose parents or legal guardians are beneficiaries of a social security scheme.

To be included, control patients (patients other than those suffering from an abdomino-pelvic tumour or malformation) must meet the following criteria:

* Patient aged between 5 months and 17 years inclusive.
* A patient being followed in the visceral surgery department for a pathology other than tumour or malformation, and requiring MRI as part of his or her diagnosis, extension assessment or monitoring.
* Patient whose parents or legal guardians have read, accepted and signed the study consent form.
* Patient whose parents or guardians are beneficiaries of a social security scheme.

Non inclusion criteria :

Patients

* Patient with a contraindication to MRI: metallic ocular foreign body, pacemaker, mechanical cardiac valve, old vascular clips on cerebral aneurysm, etc.
* Patient having participated in a therapeutic clinical trial involving a new molecule in the 30 days prior to inclusion.

Controls :

* Patient with a contraindication to MRI: ocular metallic foreign body, pacemaker, cardiac mechanical valve, old vascular clips on cerebral aneurysm, etc.
* Patient having participated in a therapeutic clinical trial involving a new molecule in the 30 days prior to inclusion.

Ages: 5 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients included in the three groups are followed in the visceral surgery department of Necker-Enfants Malades Hospital in Paris (France) for whose an MRI is required as part of diagnosis, extension assessment or monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Images produced by General Electrics' 3 Tesla MRI | through study completion, an average of 1 year
  Nerve network in areas of interest (pelvis) using tractography analysis with 3 Tesla MRI by automation of 3D imaging using images produced by General Electrics' 3 Tesla MRI. This automation will be carried out using software developed by Telecom Paristech.

SECONDARY OUTCOMES:
Post-operative consequences of surgery and/or rehabilitation treatment in patients with abdomino-pelvic tumours or pelvic malformations. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Necker enfants malades Hospital, Paris, Île-de-France Region, France